CLINICAL TRIAL: NCT03703050
Title: Phase II Trial of Nivolumab for Pediatric and Adult Relapsing/Refractory Anaplastic Large Cell Lymphoma, for Evaluation of Response in Patients With Progressive Disease Cohort 1 or as Consolidative Immunotherapy in Patients in Complete Remission After Relapse Cohort 2
Brief Title: Nivolumab for Pediatric and Adult Relapsing/Refractory ALK+, for Evaluation of Response in Patients With Progressive Disease (Cohort 1) or as Consolidative Immunotherapy in Patients in Complete Remission After Relapse (Cohort 2)
Acronym: NIVO-ALCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001447-31; 2018/2706 (Other: CSET number)
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Relapsing/Refractory ALK+ Anaplastic Large Cell Lymphoma
MeSH Terms: conditions — Recurrence | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, single arm phase II trial with 2 cohorts of ALK+ ALCL treated with nivolumab, according to patient status after previous treatment (patients in progression, into the Cohort 1; patients in CR, into the Cohort 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): Population: relapsed/refractory ALK+ ALCL with progressive disease after treatment (including chemotherapy and ALK inhibitor and/or brentuximab vedotin).
  Interventions: Drug: Nivolumab cohort 1
- Cohort 2 (Experimental): Population: patients with a relapsed/refractory ALCL, having achieved CR with a treatment including ALK-inhibitor or Brentuximab vedotin of at least 2 months and for whom HSCT is considered for their consolidation therapy. In this case, nivolumab would be considered as consolidative immunotherapy instead as HSCT.
  Interventions: Drug: Nivolumab cohort 2

INTERVENTIONS:
Drug: Nivolumab cohort 1 — Induction: nivolumab 3 mg/kg (maximal unitary dose: 240 mg) iv Q2W until CR Evaluation of response as defined below, including biopsy in case of residual masses at Week 24 Maintenance: nivolumab 3 mg/kg (maximal unitary dose: 240 mg) Q4W Total duration of treatment (induction + maintenance) = 24 months
  Other Names: OpDIVO
  Arms: Cohort 1
Drug: Nivolumab cohort 2 — Induction: nivolumab 3 mg/kg iv Q2W for 4 doses (Wk0, Wk2, Wk4 and Wk6) Maintenance: nivolumab 3 mg/kg Q4W, for 25 doses, starting at Week 8 (14 days after the last induction dose) Total duration of treatment (induction + maintenance) = 24 months
  Other Names: opdivo
  Arms: Cohort 2

SUMMARY:
Prospective, non-randomized, single arm phase II trial with 2 cohorts of ALK+ ALCL treated with nivolumab

DETAILED DESCRIPTION:
Prospective, non-randomized, single arm phase II trial with 2 cohorts of ALK+ ALCL treated with nivolumab

Cohort 1:

Population: relapsed/refractory ALK+ ALCL with progressive disease after treatment (including chemotherapy and ALK inhibitor and/or brentuximab vedotin).

Primary endpoint: ORR = best objective response rate (CR+PR) within the first 24 weeks, assessed according to adapted Lugano 2014 response criteria for Lymphoma.

Design: A one-stage phase II trial with unacceptable ORR = 40% and promising ORR = 70%. 12 eligible and evaluable patients are required.

Cohort 2 Population: patients with a relapsed/refractory ALCL, having achieved CR with a treatment including ALK-inhibitor or Brentuximab vedotin of at least 2 months and for whom HSCT is considered for their consolidation therapy. In this case, nivolumab for 24 months would be considered as consolidative immunotherapy instead as HSCT.

Primary endpoint: progression-free survival (PFS) A PFS rate ≤ 50% will be considered as unacceptable. Design: A four-stage phase II trial with unacceptable PFS rate = 50% and promising PFS rate = 75%. A maximum of twenty-six patients will be included: 4 at the 1st and 2nd stages, 8 at the 3rd stage and 10 at the 4th stage.

No more than one third of the included patients must have received more than 12 months of ALK inhibitor or brentuximab. Thus, the inclusion of these patients will be closed after 8 patients.

ELIGIBILITY:
Inclusion Criteria:

All criteria from I-1 to I-10 are required for all patients, in addition of the cohort-specific criteria

I-1. Histologically confirmed evidence of relapsed/refractory ALK+ ALCL. If biopsy could not be performed, relapsed/refractory status should be confirmed by molecular analysis whenever possible (increase of MRD quantitative PCR at 2 consecutive measures qualifying for a significant increase according to the same reference laboratory, with clinical signs and symptoms suggestive of progressing disease). In this case, relapsed/refractory status must be reviewed and confirmed by the international coordinating investigator.

I-2. Age at inclusion > 6 months

I-3. No washout needed, but patients must have recovered from acute toxic effects of all prior therapy before enrollment into the study. A short course of steroids is allowed at the beginning of Nivolumab if it is clinical indicated

I-4. Adequate organ function:

* Peripheral absolute neutrophil count (ANC) ≥750/μL in patients without bone marrow involvement and ≥500/μL in patients with bone marrow involvement (unsupported)
* Platelet count ≥75,000/μL in patients without bone marrow involvement and 50 000 in patients with bone marrow involvement (unsupported)
* Hemoglobin ≥8.0 g/dL (transfusion is allowed)
* Serum creatinine ≤1.5 x upper limit of normal (ULN) for age
* Total bilirubin ≤1.5 x ULN in patients without liver involvement and < 2.5 ULN in patients with liver involvement
* Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤3 x ULN in patients without liver involvement and < 5 ULN in patients with liver involvement
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase/SGOT ≤3 x ULN in patients without liver involvement and < 5 ULN in patients with liver involvement

I-5. Performance status: Karnofsky performance status (for patients >12 years of age) or Lansky Play score (for patients ≤12 years of age) ≥ 40%.

I-6. Able to comply with the scheduled disease management (treatment and follow-up), and with the management of toxicity

I-7. Females of childbearing potential must have a negative serum β-HCG pregnancy test within 24 hours prior to initiation of treatment. Sexually active women of childbearing potential must agree to use acceptable and appropriate contraception during the study and for at least 5 months after the last study treatment administration. Sexually active males patients must agree to use condom during the study and for at least 7 months after the last study treatment administration.

I-8. Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study-specific screening procedures are conducted according to local, regional or national guidelines.

I-9. Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.

I-10. Patients will prior allogeneic HSCT may be included if clinically indicated (see non-inclusion criteria regarding prior allogeneic HSCT). In this case, study inclusion must be confirmed by the international coordinating investigator.

Cohort 1:

For being enrolled in Cohort 1, all criteria from C1.I-1 to C1.I-2 are required, in addition of I-1 to I-10 criteria C1.I-1. Measurable progressive disease with at least one lesion measuring more than 1.5 cm and/or evaluable disease on PET-CT C1.I-2. Previous treatment including chemotherapy and ALK inhibitor or brentuximab vedotin, if available.

Cohort 2:

For being enrolled in Cohort 2, all criteria from C2.I-1 to C2.I-2 are required, in addition of I-1 to I-10 criteria C2.I-1. Complete response (disappearance of all disease except for possible detection of MRD in blood and/or bone marrow) with an on-going treatment of at least 2 months with ALK inhibitor or brentuximab vedotin, if available combined or not with chemotherapy C2.I-2. High-risk relapsed/refractory ALK+ ALCL for whom an hematopoietic stem cell transplantation is considered after CR

Exclusion Criteria:

E-1. Patients with prior allogeneic HSCT less than 3 months before study inclusion

E-2. Patients with prior allogeneic HSCT and any active graft versus host disease (GVHD) and/or any prior grade 3 or 4 GVHD according to International Bone Marrow Transplant Registry (ITBMR)

E-3. Previous organ transplantation

E-4. Significant hemophagocytosis in bone marrow, spleen, lymph nodes, or liver must be discussed with the Coordinating Sponsor before inclusion

E-5. Presence of any ≥ CTCAE grade 2 treatment-related toxicity with the exception of alopecia, fatigue and peripheral neuropathy.

E-6. History or evidence of severe uncontrolled illness that contra-indicates use of an investigational drug, or places the patient at unacceptable risk from treatment complications

E-7. History or evidence of severe acute or chronic infection unless fully healed at least four weeks prior to screening

E-8. Known human immunodeficiency virus (HIV) infection

E-9. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.

E-10. History or evidence of any auto-immune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

E-11. Subjects with another pathology requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

E-12. Known hypersensitivity to any component of the products (study drug or ingredients)

E-13. Concurrent administration of any other antitumor therapy

E-14. Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening).

E-15. Vaccinated with live attenuated vaccines within 4 weeks of the first dose of the study drug

E-16. Pregnant or breast-feeding female patient

E-17. Patient under guardianship or deprived of his liberty by a judicial or administrative decision, patients under safeguards of justice or incapable of giving its consent, patients undergoing psychiatric care under duress

E-18. Participation in another clinical study with an investigational product during the study

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 - Best objective response rate (Complete Response + Partial Response) | within the first 24 weeks
  In case of PET-positive residual masses after 24 weeks of induction treatment, a resection/biopsy must be performed by week 24. A residual mass proven to be pathologically negative for disease after resection or limited biopsy is considered as CR after discussion with the Coordinating investigator.
Cohort 2 - Progression Free Survival | up to 12 months
  PFS is defined as the time since the inclusion in the trial to the first event among relapse and death (whatever the cause of death).

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Minard, Pr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (13):
- Rigshospitalet, Copenhagen, Denmark
- France (11):
  - Gustave Roussy, Villejuif, Val De Marne
  - CHU Bordeaux Hopital Pellegrin, Bordeaux
  - CHU Bordeaux, Bordeaux
  - CHU Mondor, Créteil
  - Centre Oscar Lambret, Lille
  - Centre Léon Berard Lyon, Lyon
  - Hôpital Saint Louis, Paris
  - Hôpital Trousseau, Paris
  - CHU Toulouse Hopital des enfants, Toulouse
  - IUC Toulouse, Toulouse
  - CHU de nancy, Vandœuvre-lès-Nancy
- Women'S and Children'S Nhs Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided